CLINICAL TRIAL: NCT02906046
Title: Weight in Lower Limbs Improves Gait Ataxia Of in Machado-Joseph Disease Patients: A Randomized Crossover Trial
Brief Title: Weight in Lower Limbs Improves Gait Ataxia of in Machado-Joseph Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, giovana duarte eltz, Physiotherapist, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 989/12
Record Dates: First submitted 2016-08-24; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2013-01

CONDITIONS: Machado-Joseph Disease
Keywords: SCA 3; Ataxic Gait
MeSH Terms: conditions — Machado-Joseph Disease; Gait Ataxia | interventions — Weights and Measures

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- placebo Weight in Lower Limbs (Placebo Comparator): placebo Weight in Lower Limbs
  Interventions: Device: Weight in Lower Limbs
- 0,5 kg Weight in Lower Limbs (Other): 0,5 kg Weight in Lower Limbs
  Interventions: Device: Weight in Lower Limbs
- 1,0 kg Weight in Lower Limbs (Other): 1,0 kg Weight in Lower Limbs
  Interventions: Device: Weight in Lower Limbs

INTERVENTIONS:
Device: Weight in Lower Limbs

SUMMARY:
Few studies evaluated the efficacy of adding weights on the lower limbs in patients with ataxic disorders. There is no current evidence on which would be the most appropriate weight for use in this context. To assess progress and benefits of using this load, gait of symptomatic carriers of spinocerebellar ataxia type 3/Machado Joseph disease the objective of the study is to evaluate the gait with and without different load weights on lower limbs. Outcomes were the Scale for the Assessment and Ataxia Rating of (SARA), kinematic gait assessment by the accelerometer and gyroscope and the Patient Global Impression (PGI) about which weight they prefer for walking.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have between 18 and 65 years of age and independent gait

Exclusion Criteria:

* Were the need of assistive devices for walking ≤ 10m (such as crutches, wheelchairs and orthotics)
* Item gait of Scale for the Assessment and Rating of Ataxia (SARA)19≥, presence of other neurological disease that affect motor system
* Orthopedic impairments of lower limbs (fractures or surgeries in the past 6 months)
* Difference between the lower limbs greater than 3.0 cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Gait speed analysis [speed (mt/min) of walking for 10 meters away] | speed (mt/min) of walking for 10 meters away in 1min timeout

SECONDARY OUTCOMES:
Gait cadence analysis [cadence (steps/min) of walking for 10 meters away] | cadence (steps/min) of walking for 10 meters away in 1min timeout